CLINICAL TRIAL: NCT00406549
Title: Multi-Center Clinical Performance Evaluation of a Rapid In Vitro Diagnostic Device for Direct Detection of Staphylococcus Aureus Nasal Colonization: Comparative Analysis to Culture Screening Methods
Brief Title: Evaluation of a Diagnostic Device for Detection of Nasal Staphylococcus Aureus
Status: Completed | Type: Observational
Sponsor: Solventum US LLC (Industry)
Collaborators: 3M (Industry)
Other Study IDs: I2MS 05-010077
Record Dates: First submitted 2006-11-30; First posted 2006-12-04 (Estimated); Last update posted 2024-10-02 (Actual); Status verified 2024-09

CONDITIONS: Staphylococcus Aureus
Keywords: Staphylococcus aureus; Nasal colonization; pre-surgical patients; Sensitivity; Specificity; Nasal Staphylococcus aureus in pre-surgical patients
MeSH Terms: conditions — Staphylococcal Infections; Hypersensitivity

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
To establish the clinical test performance characteristics of sensitivity, specificity and predictive values for direct detection of nasal Staphylococcus aureus colonization against clinical microbiology laboratory culture methods.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects 18 years of age or older, male or female and from any race or culture.
2. Subjects who are ambulatory (able to walk unaided or with a cane, walker, wheelchair) on the day of their pre-operative visit for non-emergent surgery.

Exclusion Criteria:

1. Subjects who are on the nasal topical antibiotic Mupirocin (Bactroban® Nasal Ointment) within the last 4 weeks.
2. Subjects who are present at the preoperative visit with prescribed nasal medical devices (e.g. CPAP = Continuous Positive Airway Pressure or Nasal Cannula), nasal prosthetics, the wearing of nasal jewelry or trauma to the nose or anything that may inhibit sampling of the anterior nares.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2000
Dates: Start 2006-12; Study Completion 2007-03

CONTACTS AND LOCATIONS:
Overall Officials: Steve Gordon, M.D., Principal Investigator — The Cleveland Clinic
Locations (11):
- United States (8):
  - Hope Research Institute, Phoenix, Arizona
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Atlanta Institute for Medical Research, Decatur, Georgia
  - Northwestern Univesity, Chicago, Illinois
  - University of Iowa, Iowa City, Iowa
  - Johns Hopkins University, Baltimore, Maryland
  - Wake Forest University Baptist Medical Center, Winston-Salem, North Carolina
  - Cleveland Clinic Foundation, Cleveland, Ohio
- Hospital Bichat, Paris, France
- University of Muenster Hospital and Clinics, Münster, Germany
- Amphia Hospital, Breda, Netherlands